CLINICAL TRIAL: NCT04016415
Title: Decreasing Stress in Diabetes: A Randomized Controlled Trial
Brief Title: Decreasing Stress in Diabetes
Acronym: De-Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH); Rowan University (Other); West Chester University of Pennsylvania (Other); Georgetown University (Other)
Responsible Party: Principal Investigator, Nazia Raja-Khan, Associate Professor of Medicine, Obstetrics and Gynecology, and Psychiatry and Behavioral Health, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10532; 5R01DK119379 (NIH)
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Stress; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
Keywords: Stress, Psychological; Mindfulness; Meditation; Mind-Body Therapies; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Stress, Psychological | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel group two-arm trial that will determine the effects of an online 6-month Mindfulness-based stress reduction (MBSR) intervention compared to Stress Management Education (SME) (active control) on glucose control in at least 290 patients with uncontrolled diabetes. Both MBSR and SME will be delivered online by experienced instructors in a live interactive virtual classroom using videoconferencing.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI, study coordinator, and all study personnel collecting outcomes, will be blinded from the treatment assignments. Only the MBSR and SME instructors and the study personnel who schedule the classes, videorecord the classes, and code the videos will have knowledge of the assignments, and these individuals will not be involved in the collection of outcomes. Subjects will be asked to keep their treatment assignment concealed from study personnel collecting outcomes. However, complete blinding may not be possible given the nature of this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Stress Reduction (Experimental)
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Stress Management Education (Active Comparator)
  Interventions: Behavioral: Stress Management Education

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — Subjects randomized to Mindfulness-Based Stress Reduction (MBSR) will receive the 8-week University of Massachusetts Authorized MBSR curriculum followed by monthly mindfulness boosters in Months 3 to 6. The University of Massachusetts MBSR curriculum was selected for the intervention, as it is the most standardized and researched mindfulness program that has been shown to reduce psychological distress in various patient populations.
  Arms: Mindfulness Based Stress Reduction
Behavioral: Stress Management Education — Subjects randomized to Stress Management Education (SME) will receive health education on nutrition (adapted for the type 2 diabetes population), exercise as gentle stretching to match yoga in MBSR, and other general health topics that may be relevant to the type 2 diabetes population such as sleep, time management, etc. Stress Management Education does not have any mindfulness in it. Stress Management Education was specifically created as a control condition for MBSR studies so it matches MBSR for time, social support, homework, etc.
  Arms: Stress Management Education

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial (RCT) to determine the effects of an online 6-month Mindfulness-based stress reduction (MBSR) intervention compared to an active control Stress Management Education (SME) on glucose control in adults with uncontrolled type 1 or type 2 diabetes. The study will randomize at least 290 adults with uncontrolled diabetes to a 6-month MBSR intervention or SME control. Both MBSR and SME will be delivered online by experienced instructors in a live interactive virtual classroom using videoconferencing. Outcomes will be assessed at baseline, a follow-up phone call after Class #4, and study visits at 2-months (2MO) and 6-months (6MO).

DETAILED DESCRIPTION:
Specific Aims are: 1) To conduct a randomized controlled trial to determine the effects of an online 6-month Mindfulness-Based Stress Reduction (MBSR) intervention compared to an active control Stress Management Education (SME) on glucose levels in at least 290 adults with uncontrolled type 1 or type 2 diabetes. Both MBSR and SME will be delivered online by experienced instructors in a live interactive virtual classroom using videoconferencing. The primary outcome will be hemoglobin A1c (HbA1c), a measure of the average glucose level over the past 3 months. We hypothesize that between the two groups, there will be a clinically significant 0.5% absolute difference in the mean change in HbA1c from baseline to 6-months. We will also look at the 2-month HbA1c, however it may be too brief a time period to fully capture the impact of MBSR. An absolute reduction in HbA1c of 0.5% would be expected to reduce the risk of any diabetes-related complication by at least 10%. Additionally, we will assess fasting glucose as a secondary outcome as it is linked with adverse health outcomes, and can be lowered with MBSR based on our pilot study; 2) To determine the effects of online MBSR compared to SME control on psychosocial, behavioral and physiological mechanisms potentially mediating the effects of MBSR and/or SME on glucose levels in adults with uncontrolled diabetes. Secondary outcomes include: diabetes-related distress, subjective stress, craving, the impact of Coronavirus Disease 2019 (COVID-19) on subjects' lives, subject expectancy, dietary intake, physical activity, and serum hsCRP as a marker of chronic inflammation. Adverse Childhood Experiences (ACEs) will be assessed at baseline. It is hypothesized that these measures may mediate the effects of MBSR and/or SME on glucose.

The proposed study has the potential to transform current standards of care for diabetes by using a novel long-term MBSR intervention as a powerful adjunct intervention for diabetes. MBSR could impact the clinical picture of diabetes by empowering patients with skills for strengthening their own internal resources to promote self regulation and adaptive coping and reduce stress reactivity, which are all essential for implementing healthy behaviors and are expected to lead to improved glucose control and reduced risk of diabetes complications. This proposal is relevant to the mission of the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) to conduct research on diabetes to improve people's health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Men and Women
2. Age 18 years or older
3. Diagnosed with diabetes for at least one year
4. Hemoglobin A1c ≥ 7.5% within 10 weeks and 2 days (72 days) before the start of the study intervention (Orientation session)
5. High Subjective stress defined as Perceived Stress Scale-10 score ≥ 12
6. Available for the intervention sessions with reasonable certainty
7. Have a device equipped with internet connection, camera and microphone and willingness to interact with study staff and class instructors virtually/remotely via this platform
8. Must have a Primary Care Provider (PCP)
9. Must have an accessible/active personal e-mail address or be willing to obtain one for study correspondence

Exclusion Criteria:

1. Current suicidality
2. History of, or meets Mini International Neuropsychiatric Interview (MINI) structured interview criteria for, bipolar disorder, psychosis, or other significant psychopathology; Those with depression or anxiety will be allowed to participate since they are under the care of a PCP.
3. Inpatient admission for psychiatric disorder within the past two years, or ER visit for psychiatric disorder within the past 10 weeks
4. Meets MINI structured interview criteria for Alcohol Use Disorder or Substance Use Disorder (Past 12 months)
5. Inability to read, write or speak English
6. Current enrollment in a stress reduction program, or in any other investigative study
7. Previous participation in a mindfulness-based stress reduction (MBSR) course
8. Pregnant women
9. Have a household member who is currently, or was previously, assigned to study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nazia T Raja-Khan, M.D., M.S., Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available upon request approval beginning one year following the trial's initial publication date. All data requests must be submitted to the Principal Investigator (PI) in the form of a brief proposal outlining the research questions and aims, statistical analysis plan, specific measures needed, funding availability or sponsors involved (if applicable), and any other details pertaining to the proposed project. Proposals will be reviewed by the PI and relevant study team members within 3 months upon receipt.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Proposals will be reviewed and considered for approval beginning one year following the trial's initial publication date
Access Criteria: For data request proposals that receive approval, consultations will be scheduled to coordinate any relevant or applicable Institutional Review Board (IRB) considerations and/or data use agreements pertaining to the specific data requested.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from medical clinics, support groups, health fairs, StudyFinder, ResearchMatch, HealthGrades, and social media began 2/26/20 with final participant screened 1/17/24. First consent to study was 7/28/20. Type 2 diabetics were eligible for the study until 7/22/21, then expanding to all diabetics (except gestational diabetes). Eligibility was HbA1c ≥ 8 until 5/9/22, when eligible HbA1c dropped to ≥ 7.5. Final follow-up for primary outcome data collection was on 8/9/24.
Pre-assignment Details: 497 consents were signed following pre-screening at the start of the initial screening visit, reflecting n=492 unique consented individuals. Study eligibility criteria were assessed further during the screening visit and baseline visit. 183 individuals were consented but never randomized (never enrolled; n=161 ineligible at screening visit, n=1 ineligible at baseline visit, n=14 withdrew from the study, n=1 died, n=6 study team withdraws). 309 (492-183) individuals were enrolled and randomized.
Groups:
- Mindfulness Based Stress Reduction: MBSR course (Intervention) - 8-week University of Massachusetts Mindfulness-Based Stress Reduction curriculum adapted for live online delivery due to the Coronavirus Disease 2019 (COVID-19) pandemic; 1 orientation, 6 weekly classes, 1 retreat (long class session), 2 weekly classes, 4 monthly booster sessions; participants are asked to do at least 25-30 minutes of home practice homework per day for 6 days each week for the first 7 weeks following the first class. Home practice homework included mindfulness activities in accordance with the standard MBSR curriculum. Following the last weekly class, participants are encouraged to continue their home practice activities regularly on their own. Examples of MBSR activity engagement includes mindful walking, mindful yoga, mindful eating, and body scans. MBSR does not cover health education. Both arms received the following general information at their baseline visit: Two handouts from the American Diabetes Association Patient Education Library, 1) "Plan Your Portions" Diabetes Placemat and 2) "The Diabetes Advisor - Physical Activity", and three additional handouts covering 3) Hyperglycemia/Hypoglycemia, 4) Glucometer Best Practices, and 5) Blood Glucose Meter Correlation.
- Stress Management Education: SME course (Active Control) - Dr. Elizabeth Hoge's Stress Management Education program curriculum adapted for live online delivery due to the COVID-19 pandemic; 1 orientation, 6 weekly classes, 1 retreat (long class session), 2 weekly classes, 4 monthly booster sessions; participants are asked to do at least 25-30 minutes of home practice homework per day for 6 days each week for the first 7 weeks after the first class. Home practice homework included listening to excerpts of audiobooks about general stress management or nutrition facts. Following the last weekly class, participants are encouraged to continue their home practice activities regularly on their own. The SME curriculum was specifically created as a control condition for MBSR studies to parallel the intervention's structure with respect to time, schedule, social support, homework, etc. SME does not cover mindfulness. The SME program includes nutrition (adapted for individuals with diabetes), exercise as gentle stretching with Theraband to parallel the yoga component of MBSR, and other general health topics, such as sleep. Both arms received the following general information at their baseline visit: Two handouts from the American Diabetes Association Patient Education Library, 1) "Plan Your Portions" Diabetes Placemat and 2) "The Diabetes Advisor - Physical Activity", and three additional handouts covering 3) Hyperglycemia/Hypoglycemia, 4) Glucometer Best Practices, and 5) Blood Glucose Meter Correlation.
Period: Overall Study
Arm/Group | Mindfulness Based Stress Reduction | Stress Management Education
Started | 154 | 155
Attended Orientation (Began Intervention) | 147 | 149
Completed a 2-month (2MO) Visit | 123 | 124
Completed | 115 | 123
Not Completed | 39 | 32
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 6 | 2
Not completed — Physician Decision | 5 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 24 | 27
Not completed — Participant Non-Compliance: Orientation not completed prior to Class #2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants; participants age 18 or older were eligible to participate.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Stress Reduction | Stress Management Education | Total
Number analyzed (Participants) | 154 | 155 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (12.24) | 53.6 (11.67) | 54.6 (11.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 102 | 206
  Male | 50 | 53 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 15 | 21
  Not Hispanic or Latino | 147 | 138 | 285
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 19 | 40
  White | 125 | 126 | 251
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 154 | 155 | 309
Type of Diabetes [Count of Participants; unit: Participants] — Type of diabetes diagnosed for at least one year prior to trial eligibility assessment; only participants with Type 2 Diabetes were eligible to participate in the trial until 07/22/2021 (cohorts 1-4), after which time recruitment was expanded to include any type of diabetes, except gestational diabetes during pregnancy (cohorts 5-14). Therefore, this measure reflects values self-reported by participants collected during the screening visit, from the participant's electronic medical record (EMR), and/or baseline visit.
  Participants
    Type 1 | 24 | 23 | 47
    Type 2 | 127 | 128 | 255
    Latent Autoimmune Diabetes in Adults (LADA) | 0 | 3 | 3
    Diabetes due to pancreatitis or pancreatectomy (surgical removal of all or part of the pancreas) | 2 | 1 | 3
    Drug- or chemical-induced diabetes (such as with steroid use or after organ transplantation) | 1 | 0 | 1
Randomization Stratification Factor; Taking Insulin at Baseline [Count of Participants; unit: Participants] — Does the participant report currently taking any form of insulin at the time of the baseline visit prior to randomization?; self-reported by participants and verified on participant medications list by research coordinator.
  Participants
    No | 63 | 64 | 127
    Yes | 91 | 91 | 182
A1CNow® Self-Check Hemoglobin A1c (HbA1c) Home Kit Values [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] — Home Hemoglobin A1c (HbA1c) was measured using the PTS Diagnostics A1CNow® Self-Check Kit during screening and/or baseline visit (pre-randomization values). 89 values were carried forward to baseline from screening that took place within 14 days prior to baseline, and 217 values were collected at baseline. Of the n=154 participants randomized to MBSR arm, n=3 participants were missing pre-randomization values (n=2 protocol deviations - values not recollected at baseline with screening values collected > 14 days prior; n=1 protocol deviation - no pre-randomization home kit value collected). Population: Of the n=154 participants randomized to MBSR arm, n=3 participants were missing pre-randomization values (n=2 protocol deviations - values not recollected at baseline with screening values collected > 14 days prior; n=1 protocol deviation - no pre-randomization home kit value collected).
  percentage of glycated hemoglobin
    number analyzed (Participants) | 151 | 155 | 306
    (all) | 8.56 (1.3) | 8.62 (1.3) | 8.59 (1.3)
Class Cohort Number [Count of Participants; unit: Participants] — The trial enrolled 14 class cohorts. Orientation date reflects the start of the class cohort.
  Participants
    Cohort 1: Orientation Date = 09/22/2020 | 4 | 4 | 8
    Cohort 2: Orientation Date = 01/26/2021 | 4 | 2 | 6
    Cohort 3: Orientation Date = 05/06/2021 | 2 | 4 | 6
    Cohort 4: Orientation Date = 07/20/2021 | 6 | 5 | 11
    Cohort 5: Orientation Date = 09/28/2021 | 7 | 7 | 14
    Cohort 6: Orientation Date = 01/25/2022 | 8 | 10 | 18
    Cohort 7: Orientation Date = 04/19/2022 | 10 | 12 | 22
    Cohort 8: Orientation Date = 07/26/2022 | 11 | 8 | 19
    Cohort 9: Orientation Date = 10/04/2022 | 9 | 11 | 20
    Cohort 10: Orientation Date = 01/24/2023 | 19 | 21 | 40
    Cohort 11: Orientation Date = 04/18/2023 | 24 | 20 | 44
    Cohort 12: Orientation Date = 07/11/2023 | 16 | 17 | 33
    Cohort 13: Orientation Date = 09/26/2023 | 18 | 17 | 35
    Cohort 14: Orientation Date = 01/23/2024 | 16 | 17 | 33
Diabetes Distress Scale (DDS) Mean Item Score [Mean (Standard Deviation); unit: scores on a scale] — The Diabetes Distress Scale (DDS) is a 17-item survey asked on a scale from 1 ("not a problem") to 6 ("a very serious problem"), with higher scores indicating more diabetes-related distress, with a recall timeframe for the past month. The DDS Mean Item score is calculated as the average of all 17 items on the scale.
  scores on a scale | 2.50 (0.98) | 2.33 (0.89) | 2.42 (0.94)
Perceived Stress Scale-10 (PSS-10) Score [Mean (Standard Deviation); unit: scores on a scale] — The Perceived Stress Scale-10 (PSS-10) is a 10-item survey measuring subjective stress on a scale from 0 ("never") to 4 ("very often"), with a recall timeframe for the last month, collected at screening and baseline visits. The scale includes both positive and negative worded items. After reversing four positive items, the score is calculated as the sum of all 10 items (0 to 40), with higher scores indicating higher levels of perceived stress. Pts screening for cohorts 1 and 2 (until 9/3/20) were eligible if their score upon screening was at least 20; then onward, a score of at least 12.
  scores on a scale | 19.88 (6.66) | 18.39 (6.69) | 19.13 (6.71)

OUTCOME MEASURES:

1. Primary Outcome: Change in A1CNow® Self-Check Hemoglobin A1c (HbA1c) Home Kit Values From Baseline to 6-Months (6MO)
Description: Home Hemoglobin A1c (HbA1c) was measured and collected using the PTS Diagnostics A1CNow® Self-Check Kit. See Baseline Characteristics section for more details on this outcome measure. The Least Squares Means reported are model-based estimates of constructed contrasts from the linear mixed effects model further specified in the Stat Analysis results section that included fixed effects for arm, time (visit; baseline, 2MO, 6MO), the randomization stratification factor of insulin status at baseline, and the interaction between arm and time, with random effects accounting for subjects and class cohort number nested within arm, and a residual effect to account for longitudinally repeated measures over time. This outcome measure reports the difference between group arms in the change from Baseline to 6MO from this model (where all three study visit timepoints are included in the time effect).
Time Frame: Home HbA1c was collected during the screening and/or baseline visit (pre-randomization values; see Baseline Characteristics section), 2MO visit, and 6MO visit (post-randomization values). Baseline and 6MO data are reported here as the primary comparison.
Population: Following intention-to-treat (ITT) principles, all N=309 randomized participants were included in the analysis model. Therefore, the overall number of participants analyzed for this outcome remains N=309, with n=306 participants contributing values to the baseline timepoint Least Squares Mean (MBSR=151; SME=155) and n=237 contributing values to the 6MO timepoint Least Squares Mean (MBSR=114; SME=123).
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of glycated hemoglobin
Arm/Group | Mindfulness Based Stress Reduction | Stress Management Education
Number analyzed (Participants) | 154 | 155
percentage of glycated hemoglobin
  Baseline: number analyzed (Participants) | 151 | 155
  Baseline | 8.50 [8.23 to 8.77] | 8.60 [8.33 to 8.87]
  6MO: number analyzed (Participants) | 114 | 123
  6MO | 8.15 [7.85 to 8.46] | 8.24 [7.94 to 8.54]
  Change from Baseline to 6MO | -0.35 [-0.60 to -0.10] | -0.36 [-0.60 to -0.11]
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Stress Management Education; Test type: Superiority — Two-sided tests with the null hypothesis of no difference in chg from Baseline to 6MO between the two arms. The power calculation assumed a clinically meaningful diff of 0.5% and standard deviation of 0.9%. Assuming an avg class cohort size of 18 pts and an intraclass correlation coefficient estimate of 0.08 for correlation within cohorts yielded a design effect that inflated the sample size by 1+((18-1) multiplied by 0.08)=2.36. A 15% dropout rate was assumed. 145 pts per arm yielded 80% power; p = 0.96, Mixed Models Analysis — A priori significance level = 0.05; two-sided. Analyses were based upon pre-specified hypotheses, and therefore corrections for multiple testing were not made; Linear; Fixed: arm+visit[base,2MO,6MO]+insulin at base+(armXvisit interact); Random: subjects, cohort(arm); Residual: longitudinal repeated measures; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.36 to 0.34] — Change = 6MO - Baseline; Difference = SME - MBSR; Contrasts were constructed from the linear mixed model to estimate the changes

2. Secondary Outcome: Change in A1CNow® Self-Check Hemoglobin A1c (HbA1c) Home Kit Values From Baseline to 2-Months (2MO)
Description: Home Hemoglobin A1c (HbA1c) was measured and collected using the PTS Diagnostics A1CNow® Self Check Kit. See Baseline Characteristics section for more details on this outcome measure. The Least Squares Means reported are model-based estimates of constructed contrasts from the linear mixed effects model further specified in the Stat Analysis results section that included fixed effects for arm, time (visit; baseline, 2MO, 6MO), the randomization stratification factor of insulin status at baseline, and the interaction between arm and time, with random effects accounting for subjects and class cohort number nested within arm, and a residual effect to account for longitudinally repeated measures over time. This outcome measure reports the difference between group arms in the change from Baseline to 2MO from this model (where all three study visit timepoints are included in the time effect).
Time Frame: Home HbA1c was collected during the screening and/or baseline visit (pre-randomization values; see Baseline Characteristics section), 2MO visit, and 6MO visit (post-randomization values). Baseline and 2MO data are reported here as the secondary comparison
Population: Following intention-to-treat (ITT) principles, all N=309 randomized participants were included in the analysis model. Therefore, the overall number of participants analyzed for this outcome remains N=309, with n=306 participants contributing values to the baseline timepoint Least Squares Mean (MBSR=151; SME=155) and n=244 contributing values to the 2MO timepoint Least Squares Mean (MBSR=122; SME=122).
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of glycated hemoglobin
Arm/Group | Mindfulness Based Stress Reduction | Stress Management Education
Number analyzed (Participants) | 154 | 155
percentage of glycated hemoglobin
  Baseline: number analyzed (Participants) | 151 | 155
  Baseline | 8.50 [8.23 to 8.77] | 8.60 [8.33 to 8.87]
  2MO: number analyzed (Participants) | 122 | 122
  2MO | 8.27 [7.97 to 8.58] | 8.30 [8.00 to 8.61]
  Change from Baseline to 2MO | -0.23 [-0.46 to -0.01] | -0.30 [-0.52 to -0.08]
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Stress Management Education; Test type: Superiority — All hypothesis tests are two-sided (any difference), with the null hypothesis of no difference in change from Baseline to 2MO between the two arms; p = 0.68, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.38 to 0.25] — Change = 2MO - Baseline; Difference = SME - MBSR; Contrasts were constructed from the linear mixed model to estimate the changes

3. Secondary Outcome: Change in Diabetes Distress Scale (DDS) Mean Item Score From Baseline to 2-Months (2MO)
Description: The Diabetes Distress Scale (DDS) is a 17-item survey asked on a scale from 1 ("not a problem") to 6 ("a very serious problem"), with higher scores indicating more diabetes-related distress. The DDS Mean Item score is calculated as the average of all 17 items on the scale. The Least Squares Means reported are model-based estimates of constructed contrasts from the linear mixed effects model further specified in the Stat Analysis results section that included fixed effects for arm, time (visit; baseline, 2MO, 6MO), the randomization stratification factor of insulin status at baseline, and the interaction between arm and time, with random effects accounting for subjects and class cohort number nested within arm, and a residual effect to account for longitudinally repeated measures over time. This outcome measure reports the difference between group arms in the change from Baseline to 2MO from this model (where all three study visit timepoints are included in the time effect).
Time Frame: The DDS was collected during each participant's baseline, 2MO, and 6MO visit and is framed with a recall time frame of the past month. Baseline and 2MO data are reported here as the comparison for this outcome.
Population: Following intention-to-treat (ITT) principles, all N=309 randomized participants were included in the analysis model. Therefore, the overall number of participants analyzed for this outcome remains N=309, with n=309 participants contributing values to the baseline timepoint Least Squares Mean (MBSR=154; SME=155) and n=247 contributing values to the 2MO timepoint Least Squares Mean (MBSR=123; SME=124).
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Mindfulness Based Stress Reduction | Stress Management Education
Number analyzed (Participants) | 154 | 155
scores on a scale
  Baseline | 2.48 [2.34 to 2.62] | 2.31 [2.17 to 2.45]
  2MO: number analyzed (Participants) | 123 | 124
  2MO | 2.15 [2.02 to 2.29] | 2.05 [1.91 to 2.18]
  Change from Baseline to 2MO | -0.33 [-0.43 to -0.22] | -0.26 [-0.37 to -0.16]
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Stress Management Education; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.41, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.09 to 0.21] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Change in Diabetes Distress Scale (DDS) Mean Item Score From Baseline to 6-Months (6MO)
Description: The Diabetes Distress Scale (DDS) is a 17-item survey asked on a scale from 1 ("not a problem") to 6 ("a very serious problem"), with higher scores indicating more diabetes-related distress. The DDS Mean Item score is calculated as the average of all 17 items on the scale. The Least Squares Means reported are model-based estimates of constructed contrasts from the linear mixed effects model further specified in the Stat Analysis results section that included fixed effects for arm, time (visit; baseline, 2MO, 6MO), the randomization stratification factor of insulin status at baseline, and the interaction between arm and time, with random effects accounting for subjects and class cohort number nested within arm, and a residual effect to account for longitudinally repeated measures over time. This outcome measure reports the difference between group arms in the change from Baseline to 6MO from this model (where all three study visit timepoints are included in the time effect).
Time Frame: The DDS was collected during each participant's baseline, 2MO, and 6MO visit and is framed with a recall time frame of the past month. Baseline and 6MO data are reported here as the comparison for this outcome.
Population: Following intention-to-treat (ITT) principles, all N=309 randomized participants were included in the analysis model. Therefore, the overall number of participants analyzed for this outcome remains N=309, with n=309 participants contributing values to the baseline timepoint Least Squares Mean (MBSR=154; SME=155) and n=236 contributing values to the 6MO timepoint Least Squares Mean (MBSR=115; SME=121).
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Mindfulness Based Stress Reduction | Stress Management Education
Number analyzed (Participants) | 154 | 155
scores on a scale
  Baseline | 2.48 [2.34 to 2.62] | 2.31 [2.17 to 2.45]
  6MO: number analyzed (Participants) | 115 | 121
  6MO | 2.13 [1.99 to 2.27] | 1.92 [1.78 to 2.06]
  Change from Baseline to 6MO | -0.34 [-0.47 to -0.22] | -0.39 [-0.51 to -0.27]
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Stress Management Education; Test type: Superiority — All hypothesis tests are two-sided (any difference), with the null hypothesis of no difference in change from Baseline to 6MO between the two arms; p = 0.59, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.22 to 0.12] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change in Perceived Stress Scale-10 (PSS-10) Score From Baseline to 2-Months (2MO)
Description: PSS-10 is a 10-item survey that includes both positive and negative phrased items on a scale of 0-4. After reversing 4 positive items, the summative score ranges from 0-40, where higher values indicate higher levels of perceived stress, with a recall time frame for the last month. The Least Squares Means reported are model-based estimates of constructed contrasts from the linear mixed effects model further specified in the Stat Analysis results section that included fixed effects for arm, time (visit; baseline, 2MO, 6MO), the randomization stratification factor of insulin status at baseline, and the interaction between arm and time, with random effects accounting for subjects and class cohort number nested within arm, and a residual effect to account for longitudinally repeated measures over time. This outcome measure reports the difference between group arms in the change from Baseline to 2MO from this model (where all three study visit timepoints are included in the time effect).
Time Frame: PSS-10 was assessed at screening, baseline (pre-randomization), 2MO, and 6MO visits. Baseline and 2MO data are presented here as the comparison for this outcome.
Population: Following intention-to-treat (ITT) principles, all N=309 randomized participants were included in the analysis model. Therefore, the overall number of participants analyzed for this outcome remains N=309, with n=309 participants contributing values to the baseline timepoint Least Squares Mean (MBSR=154; SME=155) and n=246 contributing values to the 2MO timepoint Least Squares Mean (MBSR=123; SME=123).
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Mindfulness Based Stress Reduction | Stress Management Education
Number analyzed (Participants) | 154 | 155
scores on a scale
  Baseline | 19.85 [18.61 to 21.09] | 18.18 [16.95 to 19.41]
  2MO: number analyzed (Participants) | 123 | 123
  2MO | 16.65 [15.35 to 17.95] | 16.55 [15.25 to 17.85]
  Change from Baseline to 2MO | -3.20 [-4.26 to -2.14] | -1.63 [-2.69 to -0.58]
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Stress Management Education; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.04, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.57, 95% CI 2-sided [0.07 to 3.06] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Change in Perceived Stress Scale-10 (PSS-10) Score From Baseline to 6-Months (6MO)
Description: PSS-10 is a 10-item survey that includes both positive and negative phrased items on a scale of 0-4. After reversing 4 positive items, the summative score ranges from 0-40, where higher values indicate higher levels of perceived stress, with a recall time frame for the last month. The Least Squares Means reported are model-based estimates of constructed contrasts from the linear mixed effects model further specified in the Stat Analysis results section that included fixed effects for arm, time (visit; baseline, 2MO, 6MO), the randomization stratification factor of insulin status at baseline, and the interaction between arm and time, with random effects accounting for subjects and class cohort number nested within arm, and a residual effect to account for longitudinally repeated measures over time. This outcome measure reports the difference between group arms in the change from Baseline to 6MO from this model (where all three study visit timepoints are included in the time effect).
Time Frame: PSS-10 was assessed at screening, baseline (pre-randomization), 2MO, and 6MO visits. Baseline and 6MO data are presented here as the comparison for this outcome.
Population: Following intention-to-treat (ITT) principles, all N=309 randomized participants were included in the analysis model. Therefore, the overall number of participants analyzed for this outcome remains N=309, with n=309 participants contributing values to the baseline timepoint Least Squares Mean (MBSR=154; SME=155) and n=238 contributing values to the 6MO timepoint Least Squares Mean (MBSR=115; SME=123).
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Mindfulness Based Stress Reduction | Stress Management Education
Number analyzed (Participants) | 154 | 155
scores on a scale
  Baseline | 19.85 [18.61 to 21.09] | 18.18 [16.95 to 19.41]
  6MO: number analyzed (Participants) | 115 | 123
  6MO | 17.04 [15.64 to 18.45] | 16.21 [14.82 to 17.59]
  Change from Baseline to 6MO | -2.81 [-3.93 to -1.68] | -1.98 [-3.07 to -0.88]
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Stress Management Education; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.30, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.83, 95% CI 2-sided [-0.74 to 2.40] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from consent through end of trial for each individual (up to roughly 6 months after orientation). Adverse events were followed until resolution/stabilization or until end of trial.
Description: All Serious Adverse Events (SAEs) are reported here for all consenting individuals. Adverse Events (AEs) were regularly solicited at baseline, 4-wk call, 2MO, and 6MO visits via systematic open-ended check-ins ("Have there been any changes to your health since the last visit?") and questionnaires (e.g. Hypoglycemia Survey) through self-report. Self-initiated reporting of AEs between visits was encouraged. Efforts were made to obtain supporting documentation from medical records as needed.
Groups:
- Consented - Not Randomized: Individuals who consented to the trial but were not randomized to a study group arm.
Arm/Group | Mindfulness Based Stress Reduction | Stress Management Education | Consented - Not Randomized
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/155 | 1/183
Serious Adverse Events (participants affected / at risk) | 15/154 | 18/155 | 1/183
Other Adverse Events (participants affected / at risk) | 43/154 | 46/155 | 0/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Based Stress Reduction (N=154) | Stress Management Education (N=155) | Consented - Not Randomized (N=183)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Conduction Disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Bone Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 3 (3) | 2 (7) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 5 (9) | 5 (9) | 0 (0)
Rotator Cuff Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cutaneous T-cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal Ideations (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Renal Calculi (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event subacute thrombosis right leg bypass graft (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness Based Stress Reduction (N=154) | Stress Management Education (N=155) | Consented - Not Randomized (N=183)
Hypoglycemia (Metabolism and nutrition disorders) | 33 (56) | 32 (59) | 0 (0)
COVID-19 (Infections and infestations) | 12 (12) | 17 (17) | 0 (0)

LIMITATIONS AND CAVEATS:
The study could not be conducted without participant awareness of their randomly assigned course. Course cohorts were variable in size. SME course cohorts were taught by several different instructors throughout the duration of the trial. The COVID-19 pandemic may have impacted participant stress. HbA1c was measured using home kits. Study visits were conducted remotely, and surveys were completed electronically, therefore biasing the study sample towards more technologically capable participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT04016415/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/15/NCT04016415/ICF_001.pdf